CLINICAL TRIAL: NCT02123420
Title: Platform Switching vs Regular Platform Implants. One Year Results From a RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Responsible Party: Principal Investigator, Silvio Mario Meloni, DDS, Phd, MS, Università degli Studi di Sassari
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PS vs RP
Record Dates: First submitted 2014-04-16; First posted 2014-04-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Missing Teeth
Keywords: Platform Switching vs Regular Platform
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Implant outcome (Other): This study was designed as a randomised, controlled, split-mouth trial. all enrolled patients needed single bilateral fixed implant-supported prosthesis in molar area.
  A total of 18 consecutive patients were enrolled. In each eligible patient, the right molar was randomly selected to receive either Nobel Replace Tapered Groovy implant; (Nobel Biocare®, Goteborg, Sweden) with Platform Switching (PS) or Regular Platform (RP)
  Interventions: Device: Nobel Replace Tapered Groovy implant; (Nobel Biocare®, Sweden)
- Implant outome (Other): This study was designed as a randomised, controlled, split-mouth trial. all enrolled patients needed single bilateral fixed implant-supported prosthesis in molar area.
  A total of 18 consecutive patients were enrolled. In each eligible patient, the left molar was randomly selected to receive either Nobel Replace Tapered Groovy implant; (Nobel Biocare®, Goteborg, Sweden) with Platform Switching (PS) or Regular Platform (RP)
  Interventions: Device: Nobel Replace Tapered Groovy implant; (Nobel Biocare®, Sweden)

INTERVENTIONS:
Device: Nobel Replace Tapered Groovy implant; (Nobel Biocare®, Sweden) — Both sites received tapered implants with an anodised surface, one site received: Nobel Replace Tapered Groovy PS implant; (Nobel Biocare, Goteborg, Sweden), with diameters of 4.3 or 5.0 mm and lengths of 10 or 8 mm, (PS group), the contralateral site received Nobel Replace Tapered Groovy implant with Replace Select connection with diameters of 4.3 or 5.0 mm and lengths of 10 or 8 mm, (RP group).
  Healing abutments were connected to implants at the same time of surgery , then flaps were sutured with Vicryl 4.0 sutures (Vicryl, Ethicon J&J International, St-Stevens-Woluwe, Belgium).
  Other Names: Nobel Replace Tapered Groovy PS implant; (Nobel Biocare®, Sweden); Nobel Replace Tapered Groovy implant with Replace Select connection (Nobel Biocare®, Sweden)

SUMMARY:
The present study tested the hypothesis that Platform Switching (PS) and Regular Platform (RP) implants would have different outcomes in the bilateral single tooth replacements against the alternative hypothesis of no difference.

DETAILED DESCRIPTION:
This study was designed as a randomised, controlled, split-mouth trial. Eighteen patients, with bilaterally missing single bicuspid or molar had one of the sites to be restored randomly assigned to be treated according to the platform-switching concept with (PS group), or with matching implant-abutment diameters, (RP group). A total of 36 implants, (18 Nobel Replace Tapered Groovy PS, 18 Nobel Replace Tapered Groovy), were bilaterally installed. All the implants were inserted with an insertion torque between 35 and 45 Ncm, in healed healthy bone and the healing abutment was connected at the same time. Both implants were delayed loaded with screw retained temporary crowns 3 months after implant insertion and with screw retained definitive crowns 2 months later. Outcome measures were implant survival, biological and prosthetic complications, radiographic marginal bone-level changes, soft tissue parameters (PPD and BOP). Clinical data were collected at baseline 6 and 12 months. Statistical analyses were conducted using computational program SAS (version 9.2), with 1-away ANOVA and F-test. Statistical significance was tested at the 0.05 probability level, and all values were presented as mean and standard deviation with 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* need for single bilateral fixed implant-supported prosthesis in molar area
* stable interocclusal contacts
* ≥18 years of age
* provided written informed consent
* residual bone height ≥10 mm
* residual bone thickness ≥6 mm with at least 5 mm of keratinised gingiva crestally

Exclusion Criteria:

* general contraindications to implant surgery
* lack of occluding dentition in the area intended for immediate loading
* periodontitis
* bruxism
* immunosuppression
* previous history of irradiation of the head and neck area
* uncontrolled diabetes
* heavy smoker (>10 cigarettes/day)
* poor oral hygiene
* current or past treatment with bisphosphonates
* substance abuse
* psychiatric disorder
* inability to complete follow-up ≥1 year
* lactation
* implant insertion torque less than 35 Ncm

Ages: 24 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Implant Survival | Up to 12 months
  implant survival: The removal of implants was dictated by instability, progressive marginal bone loss, infection or implant fracture.

SECONDARY OUTCOMES:
Change in marginal bone levels | Baseline, 12 months
  Marginal bone levels: Peri-implant marginal bone levels were evaluated on intraoral digital radiographs taken with the parallel technique at the time of implant placement, at 6 months and 12 months.
  If radiographs were inconclusive, they were repeated. A blinded radiologist (F.G.), unaffiliated with the study centre, interpreted all radiographs. The distances from the mesial and distal interproximal bone to the reference point (the horizontal interface between the implant and abutment) were measured with a software measurement tool (NIH Scion Image programme version 4.0.2, Frederick, MD, USA) calibrated against the space between two threads to the nearest 0.1 mm, and the mean of these two measurements was calculated for each implant. The measurements were recorded with reference to the implant axis.

OTHER OUTCOMES:
Change in peri-implant mucosal response parameters. | Baseline, 12 months
  Peri-implant mucosal response: Probing pocket depth (PPD) and bleeding on probing (BOP) were measured by a blinded operator (A.D.) with a periodontal probe (PCP-UNC 15, Hu-Friedy Manufacturing, Chicago, IL, USA) at 6 and 12 months. Three vestibular and 3 lingual values were collected for every implant by the same dentist.